CLINICAL TRIAL: NCT03443700
Title: Randomized Controlled Trial on Rehabilitation Training With a Robotic Anthropomorphic Exoskeleton in Patients With Motor Incomplete Spinal Cord Injury: Clinical Outcomes and Cortical Plasticity Indicators
Brief Title: Randomized Controlled Trial on Robotic Exoskeleton in Spinal Cord Injury: Clinical Outcomes and Cortical Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: IRCCS Institute of Neurological Sciences of Bologna (Italy) (Unknown); Department of Biomedical and Neuromotor Sciences of the University of Bologna (Italy) (Unknown); Montecatone Rehabilitation Institute S.p.A., Imola (Italy) (Unknown); IRCCS Fondazione S. Lucia, Roma (Italy) (Unknown); IRCCS Fondazione Ospedale S. Camillo, Venezia (Italy) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE-19072; 347-2019-DISP-AUSLBO (Other: CE AVEC)
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; gait; incomplete motor SCI; robotic gait training; locomotor training; walking training; rehabilitation; exoskeleton; EKSO; EKSO-GT; neuroplasticity; brain cortical plasticity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Because of the use of an evident Medical Device (exoskeleton), enrolled subjects cannot be blind about their assignment group, however objective and standardized clinical measure scales will be employed; moreover, assessments (also neurophysiological and neuroimaging ones) will be conducted by blind experts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- sLT (Active Comparator): Standard neurorehabilitation locomotor training during the whole study period (8 weeks).
  Interventions: Procedure: Standard neurorehabilitation locomotor training
- sLT + EX-T (Experimental): Standard neurorehabilitation locomotor training (sLT) during the whole study period (8 weeks), plus a training with a new-generation robotic anthropomorphic exoskeleton (EKSO-GT locomotor training) during the first 4 study weeks.
  Interventions: Device: EKSO-GT; Procedure: Standard neurorehabilitation locomotor training

INTERVENTIONS:
Device: EKSO-GT — Each rehabilitation session with EKSO-GT will last (operating time) 30-40 minutes. Such training will be carried out for 3 sessions per week, during the first 4 consecutive weeks of the study period (i.e. 12 total sessions per patient).
  Arms: sLT + EX-T
Procedure: Standard neurorehabilitation locomotor training — Neurorehabilitation locomotor training will be performed according to standardized protocols shared within the scientific community, during the whole 8-week study period, 5 times per week, twice a day, for a total of about 2,5 hours per day.

SUMMARY:
The recent introduction of robotics for locomotor training in paraplegic patients, and in particular the use of anthropomorphic exoskeletons, has opened new frontiers in rehabilitation. Existing literature, though encouraging, is still scarce and studies demonstrating efficacy are highly heterogeneous and have a small sample size. Evidence is also needed about cortical plasticity after SCI, in conjunction with the use of innovative rehabilitation devices, through indicators like neurophysiological and neuroradiological markers, as the knowledge of such mechanisms is crucial to improve clinical outcomes. Cortical circuits controlling prosthetic devices are different from those controlling normal parts of the body and remodeling mechanisms following prosthetic use have been documented, but in conditions other than SCI.

The aims of this randomized controlled trial, with a 2-arm parallel-group design, are:

1. to evaluate and quantify the efficacy of locomotor rehabilitation with a robotic anthropomorphic exoskeleton (EKSO-GT) in terms of clinical and functional outcomes, and the persistence of such efficacy;
2. to investigate the presence and persistence of brain neuronal plasticity and cortical remodeling mechanisms underlying the robotic rehabilitation approach.

Fifty patients will be recruited and randomly assigned to 2 treatment arms. Both groups will follow a program of standard locomotor rehabilitation for 8 weeks. One group will also undergo an overground locomotor training with the EKSO-GT during the first 4 weeks.

DETAILED DESCRIPTION:
The increasing incidence of incomplete Spinal Cord Injury (SCI) has raised new rehabilitation challenges. Recovery of walking is one of the top priorities in SCI persons and growing efforts have been pursued aimed at identifying effective alternative techniques for improving gait performance.

Standard rehabilitation approach has been so far the most widely used, but the recent introduction of anthropomorphic exoskeletons may open new frontiers in the field. Anthropomorphic exoskeletons have been developed to assist SCI patients with mobility, but there is also a certain optimism that they may have potentialities to improve walking patterns of incomplete SCI persons after a rehabilitation period with such devices is terminated. So far, however, while different systematic reviews and meta-analyses have reported on the safety of the training with such exoskeletons, there are no significant Fiftystudies on its efficacy. Along with this, central mechanisms underlying the anatomical and functional changes induced by these approaches have never been investigated in SCI.

This longitudinal randomized controlled trial, with a 2-arm parallel group design, aims at evaluating the efficacy of the training with an anthropomorphic, robotized exoskeleton (EKSO-GT, by Ekso Bionics), as "add-on" to the standard locomotor rehabilitation, in improving walking performance, when compared to the standard locomotor rehabilitation alone, in a population of patients with non-acute motor incomplete SCI. Along with this and other clinical outcomes, neurophysiological and structural markers of Central Nervous System (CNS) plasticity will be explored, aimed at capturing mechanisms underlying how anthropomorphic exoskeletons affect CNS plasticity.

Fifty patients will be recruited in 3 Italian rehabilitation hospitals setting and assigned to 2 groups, with an allocation ratio of 1:1, through a block randomization approach. One group will perform a 4-week standard locomotor training (sLT) alone, while the other will perform a 4-week period sLT plus a training with the EKSO-GT (sLT + EX-T). Afterwards, both groups will undergo a further 4-week sLT alone.

Patients will be evaluated at several time points (always when the exoskeleton is not worn): clinical outcomes will be assessed by means of clinical examinations, standardized tests and validated scales; neurophysiological modulations will be evaluated by means of paired Motor and Sensory Evoked Potentials and a study of Electroencephalographic (EEG) slow waves oscillations and signal coherence during sleep; anatomical and structural cortical modifications will be studied with brain functional Magnetic Resonance Imaging (fMRI).

It is expected that the overground locomotor training with a new-generation exoskeleton, as "add-on" to standard locomotor training, can further improve clinical outcomes (especially walking performance) in the studied population, and that such clinical improvements are underlined by mechanisms modulating synaptic plasticity occurring also at the CNS level.

ELIGIBILITY:
Inclusion Criteria:

* SCI due to traumatic or vascular etiology;
* Incomplete motor SCI (C or D in ASIA Impairment Scale);
* T1-L1 (included) neurological level;
* 1-5 years since injury;
* Functional gait ability (also with braces or orthoses);
* Sufficient Range of Motion (ROM) of lower limbs joints to achieve a reciprocal gait pattern and allow transition from sitting to vertical position;
* Stable clinical conditions;
* Minimum height of 157 cm;
* Maximum height of 188 cm;
* Maximum weight of 100 Kg;
* Maximum intertrochanteric distance of 46 cm;
* Cognitive integrity and full collaboration of the subject.
* Specific research informed consent signed.

Exclusion Criteria:

* Intensive walking rehabilitation training undergone in the last 3 months;
* Previous use of a robotic exoskeleton;
* Instability or major deformity of the spine;
* Lower limbs joints instability;
* Indication to spinal orthosis;
* Uncontrolled spasticity (score > 3 of the Modified Ashworth Scale) in the majority of the muscle groups of the lower limbs;
* History of traumatic brain injury;
* Recent significant bone fractures, traumatic and/or pathological for the required training;
* Presence of neurogenic paraosteoarthropathies (POAN) at the onset or phlogistic phase;
* Discrepancy in femurs length (> 1.3 cm) and legs length (> 1.9 cm);
* Symptomatic orthostatic hypotension;
* Severe and recurrent uncontrolled autonomic dysreflexia;
* Cardiopulmonary comorbidities limiting physical effort;
* Skin lesions that can interfere with the study rehabilitation trainings;
* Documented psychiatric pathology;
* Contraindications to fMRI and polygraphic EEG execution;
* Contraindications to TMS;
* Ongoing pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in walking performance | Baseline (initial visit post-randomization); week 4
  10-meter walk test

SECONDARY OUTCOMES:
Change in walking performance | Baseline (initial visit post-randomization); week 8
  10-meter walk test
Change in walking endurance | Baseline (initial visit post-randomization); week 4; week 8
  6-minute walk test
Change in functional walking capacity | Baseline (initial visit post-randomization); week 4; week 8
  Walking Index for Spinal Cord Injury II (WISCI II)
Change in spasticity | Baseline (initial visit post-randomization); week 4; week 8
  Modified Ashworth Scale
Change in pain | Baseline (initial visit post-randomization); every day, twice a day for the whole study period; overall appraisal at week 4 and week 8
  Numeric Rating Scale (NRS)
Change in mood state | Baseline (initial visit post-randomization); week 4; week 8
  Profile of Mood States questionnaire (POMS)
Change in lower limbs muscle strength | Baseline (initial visit post-randomization); week 4; week 8
  Lower Extremity Motor Score (LEMS) of the American Spinal Injury Association (ASIA) Impairment Scale
Change in lower limbs muscle activation pattern | Baseline (initial visit post-randomization); week 4; week 8
  Gait Dynamic Electromyography (DEMG)
Change in entity of neuronal plasticity and cortical remodelling of motor cortical areas | Baseline (initial visit post-randomization); after the first locomotor training session; week 4; week 8
  Change in short-term intracortical inhibition through Motor Evoked Potentials (PEMs) elicited by Transcranial Magnetic Stimulation (TMS)
Change in entity of neuronal plasticity and cortical remodelling of sensory cortical areas | Baseline (initial visit post-randomization); after the first locomotor training session; week 4; week 8
  Somatosensory Evoked Potentials (SSEs) at cortical level
Change in synaptic potentiation (neuroprosthetic learning) | Baseline (initial visit post-randomization); after the first locomotor training session; week 4
  Analysis of slow-wave oscillations with Electroencephalographic (EEG) polysomnography (PSG)
Change in synaptic potentiation (neuroprosthetic learning) | Baseline (initial visit post-randomization); after the first locomotor training session; week 4
  Analysis of EEG coherence signal
Change in brain anatomy and cortical structure | Baseline (initial visit post-randomization); week 4; week 8
  Functional Magnetic Resonance Imaging (fMRI)
Evaluation of patient's satisfaction for the training received | Week 4
  Ad-hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elena Antelmi, MD, Principal Investigator — IRCCS - ISNB
Locations (1):
- Azienda USL di Bologna, Istituto delle Scienze Neurologiche di Bologna (IRCCS ISNB), Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided